CLINICAL TRIAL: NCT03791398
Title: BrUOG 379: A Phase Ib/II Single Arm Study of ONC201 Plus Nivolumab in Microsatellite Stable (MSS) Metastatic Colorectal Cancer (mCRC) Patients
Brief Title: BrUOG 379 Phase Ib/II Trial ONC201 + Nivolumab in MSS mCRC
Acronym: 379
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); Bristol-Myers Squibb (Industry); Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 379
Record Dates: First submitted 2018-12-26; First posted 2019-01-02 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic; colorectal cancer; colon cancer; microsatellite stable
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms | interventions — TIC10 compound; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a single arm study of de-escalating arms to determine the MTD and then expand the trial.It is not randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ONC201 Level 1 (Starting Dose Level) (Experimental): 625mg ONC201 Cycle 1 Day -7 dose then once week
  Interventions: Drug: Dose level 1 ONC201 625mg
- ONC201 Level 2 (Experimental): 500 mg ONC201 Cycle 1 Day -7 dose then once week
  Interventions: Drug: Dose level 2 ONC201 500mg
- ONC201 Level 3 (Experimental): 375 mg ONC201 Cycle 1 Day -7 dose then once week
  Interventions: Drug: Dose level 3 ONC201 375mg
- Nivolumab (Experimental): 240mg IV flat dose q 2 weeks
  Interventions: Drug: Dose level 1 ONC201 625mg; Drug: Dose level 2 ONC201 500mg; Drug: Dose level 3 ONC201 375mg

INTERVENTIONS:
Drug: Dose level 1 ONC201 625mg — ONC201 625mg + Nivolumab 240mg IV flat dose
  Other Names: ONC201 + Nivolumab
  Arms: Nivolumab; ONC201 Level 1 (Starting Dose Level)
Drug: Dose level 2 ONC201 500mg — ONC201 500mg + Nivolumab 240mg IV flat dose
  Other Names: ONC201 + Nivolumab
  Arms: Nivolumab; ONC201 Level 2
Drug: Dose level 3 ONC201 375mg — ONC201 375mg + Nivolumab 240mg IV flat dose
  Other Names: ONC201 + Nivolumab
  Arms: Nivolumab; ONC201 Level 3

SUMMARY:
This is a single arm Phase Ib/II, open label, safety, pharmacokinetic, pharmacodynamics and efficacy study of ONC201 in combination with Opdivo (Nivolumab) in adult patients with metastatic colorectal cancer, for whom no standard therapy is available. This study will enroll adult patients with metastatic colorectal cancer who progressed after at least two lines of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically/cytologically -confirmed primary colorectal tumor, with confirmation of being microsatellite stable.
2. Radiographic or clinical evidence of metastatic disease that has progressed after at least 2 prior regimens. Prior bevacizumab, cetuximab, trifluridine and tipiracil , or regorafenib is allowed, prior FOLFIRI and FOLFOX treatment is required. (Treatment with a FOLFIRINOX regimen will count as 2 regimens). Prior treatment does not have to have been in the metastatic setting.
3. Patients must have measurable disease by RECIST criteria
4. All patients must have a tumor(s) located in an area that that can be biopsied as confirmed by treating physician
5. All patients must submit representative tissue from their malignancy if it is confirmed there is enough tissue from prior surgery or most recent biopsy.
6. All previous therapies for cancer, including radiotherapy, major surgery and investigational therapies must be discontinued for ≥ 14 days before the first dose of ONC201
7. All clinically significant adverse events related to any prior therapy must have resolved to Grade ≤ 1 Common Terminology Criteria for Adverse Events (CTCAE v5.0), except alopecia or parameters defined in this eligibility list.
8. Age ≥ 18 years.
9. ECOG performance status ≤ 2.
10. Adequate organ and marrow function as defined below:

    1. Absolute neutrophil count ≥1,000/mm3 without growth factor use ≤ 7 days prior to treatment
    2. Platelets ≥75,000/mm3 without platelet transfusion ≤ 7 days prior to treatment
    3. Hemoglobin>8.0 mg/dL without red blood cell transfusion ≤ 7 days prior to treatment
    4. Total serum bilirubin<1.5 X upper limit of normal (ULN)
    5. AST (SGOT)/ALT (SGPT)≤2 X ULN; ≤ 5 X ULN if liver dysfunction is felt to be secondary to tumor burden within 14 days prior to treatment, Serum creatinine ≤ 1.5 X ULN (OR creatinine clearance ≥ 60 mL/min/1.73 m2) within 14 days prior to treatment
    6. Serum or urine pregnancy test (for females of childbearing potential) negative ≤7 days of treatment
11. Ability to understand and the willingness to sign a written informed consent document and comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
12. Female patients of child-bearing potential must be practicing an effective form of contraception from the time of informed consent and for the duration of the study treatment through 5 months after the last dose of drug (ONC201 or Nivolumab, whichever is administered last). The decision of effective contraception will be based on the judgment of the principal investigator or a designated associate.
13. Male patients must be surgically sterile (provide date of surgery) or must agree to use effective contraception from the time of informed consent and for the duration of the study treatment through 7 months after the last dose of drug (ONC201 or Nivolumab, whichever is administered last). The decision of effective contraception will be based on the judgment of the principal investigator or a designated associate.
14. Patients must agree to the required tumor biopsies to enroll in the trial.

Exclusion Criteria:

1. Patients with symptomatic brain metastases are excluded. Patients with asymptomatic and treated CNS metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases > 28 days prior to registration, including radiotherapy or surgery. Steroids for the treatment of brain metastasis are not permitted.
2. Patients with prior treatment with ONC201 will be excluded
3. Active inflammatory gastrointestinal disease such as severe chronic diarrhea (unless related to underlying malignancy), gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study registration. Gastroesophageal reflux disease under controlled treatment with proton pump inhibitors is allowed.
4. Pregnant or breast feeding.
5. Current active treatment in another clinical study (treatment trial) within 14 days of D-7.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics, hepatitis, active rheumatologic or collagen vascular disease, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness. (testing is not required for eligibility).
8. Any of the following in the previous 3 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism as defined by treating physician.
9. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the patient inappropriate for entry into the study.
10. Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
11. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of day 1 of treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
12. Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer are excluded if there is any evidence of other malignancy being present within the last three years (2 years for invasive breast cancer). However, patients with a malignancy that is non-likely to require treatment, as per the treating physician, in the next 2 years, such as a completely resected, early stage breast cancer, or other malignancies treated with curative intent are eligible. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
13. Prior treatment with immunotherapy for any cancer, including immune checkpoint inhibitors or anti-CTLA4 agents
14. Participants who have received a live / attenuated vaccine within 30 days of first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lifespan Cancer Institute: The Miriam and Rhode Island Hospitals, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ONC201 Level 1 (Starting Dose Level) | ONC201 Level 2 | ONC201 Level 3
Started | 13 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Progression of Disease Under Study | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled to dose level 2 or 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | ONC201 Level 1 (Starting Dose Level) | ONC201 Level 2 | ONC201 Level 3 | Total
Number analyzed (Participants) | 13 | 0 | 0 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 8 |  |  | 8
  >=65 years | 5 |  |  | 5
Age, Continuous [Mean (Full Range); unit: years] | 60 [34 to 84] |  |  | 60 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 |  |  | 8
  Male | 5 |  |  | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 1
  Not Hispanic or Latino | 12 |  |  | 12
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 3 |  |  | 3
  White | 9 |  |  | 9
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 |  |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of ONC201 With Nivolumab for Phase II
Time Frame: Cycle 1 (each cycle is approximately 4 weeks) through pre-dosing cycle 2, approximately 1 month
Measure: Number; unit: mg
Arm/Group | ONC201 Level 1 (Starting Dose Level)
Number analyzed (Participants) | 11
mg | 625

2. Primary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From start of protocol therapy until death or progression, a maximum of 6 months from end of therapy.
Measure: Mean (Full Range); unit: days
Arm/Group | ONC201 Level 1 (Starting Dose Level)
Number analyzed (Participants) | 11
days | 58 [9 to 97]

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time a signed and dated ICF is obtained until 100 days (+1 week) after the last treatment (Nivolumab or ONC201, whichever is last), or until the subject withdraws consent from study participation or at the time patient becomes a screen failure, whichever occurs first. An average of 6 months.
Arm/Group | ONC201 Level 1 (Starting Dose Level)
All-Cause Mortality (participants affected / at risk) | 11/13
Serious Adverse Events (participants affected / at risk) | 10/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONC201 Level 1 (Starting Dose Level) (N=13)
Small intestinal obstruction (Gastrointestinal disorders) | 4
Blood bilirubin increased (Investigations) | 1
Fungemia (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 8
Hematuria (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Abdominal infection (Infections and infestations) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Endoscopic retrograde cholangiopancreatography (Surgical and medical procedures) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Muscle weakness right-sided (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONC201 Level 1 (Starting Dose Level) (N=13)
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 5
Gastritis (Gastrointestinal disorders) | 1
Abdominal cramping (Gastrointestinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Thyroid stimulating hormone increased (Investigations) | 2
Vomiting (Gastrointestinal disorders) | 1
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT03791398/Prot_SAP_ICF_000.pdf